CLINICAL TRIAL: NCT07234201
Title: Designing a Virtual Reality Intervention to Improve Physical and Psychological Health in Intensive Care Units
Brief Title: Virtual Reality Use for ICU Mobility
Acronym: GAMERS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PRO00116448_1
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Intensive Care Unit ICU

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Standard mobility care
- VR intervention (Other): Virtual Reality
  Interventions: Other: Nurse driven virtual reality mobility session

INTERVENTIONS:
Other: Nurse driven virtual reality mobility session — Participants will use the virtual reality device to play the game that will facilitate movement of arms, shoulders and trunk to music, similar to dancing or Tai-Chi.
  Arms: VR intervention

SUMMARY:
The purpose of this study is to explore if Virtual Reality (VR) helps patients in the Intensive Care Unit (ICU) move more and feel better.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Adults age 18 or greater
* ICU stay greater or equal to 3 days
* Limited mobility

Exclusion Criteria:

* Pregnancy
* Special enteric contact isolation
* Blindness
* History of seizure or vertigo
* Intubated and sedated
* ICU delirium

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Increased Mobility | 10 days or ICU discharge, which ever comes first

SECONDARY OUTCOMES:
Number of participants with Improved psychosocial well-being | 10 days or ICU discharge, which ever comes first

CONTACTS AND LOCATIONS:
Overall Officials: Anna Mall, Principal Investigator — Duke University
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No